CLINICAL TRIAL: NCT01983722
Title: Treatment Plan to Provide Expanded Access to Stiripentol for Patients With Dravet Syndrome
Status: Approved for marketing | Type: Expanded Access
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-5518
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Dravet Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — stiripentol

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Stiripentol

SUMMARY:
Expanded access to Stiripentol for patients with Dravet Syndrome.

DETAILED DESCRIPTION:
This is a treatment plan, and therefore patients will be monitored according to clinical standard of care.

ELIGIBILITY:
Inclusion Criteria:

* 6 months and older
* Diagnosis of Dravet Syndrome with intractable seizures

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients
* Past history of psychoses in the form of episodes of delirium
* Impaired hepatic and/or renal function, defined as creatinine >2 and/or transaminase >4xULN

Min Age: 6 Months | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States